CLINICAL TRIAL: NCT02137850
Title: An Open-label Single-arm Multicentre Non-controlled Phase 3a Trial Investigating Safety and Efficacy of N8-GP in Prophylaxis and Treatment of Bleeding Episodes in Previously Untreated Paediatric Patients With Severe Haemophilia A
Brief Title: Safety and Efficacy of Turoctocog Alfa Pegol (N8-GP) in Previously Untreated Patients With Haemophilia A
Acronym: pathfinder™6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7088-3908; 2013-004025-88 (EudraCT Number); U1111-1148-1897 (Other: WHO); REec-2014-0898 (Registry Identifier: Spanish Register of Clinical Studies (REec)); JapicCTI-142577 (Other: JAPIC)
Record Dates: First submitted 2014-03-28; First posted 2014-05-14 (Estimated); Results first posted 2024-10-31 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 50 EDs (exposure days) (Experimental)
  Interventions: Drug: turoctocog alfa pegol

INTERVENTIONS:
Drug: turoctocog alfa pegol — For intravenous (i.v.) injection. Frequency and dosage (20-75 U/kg) dependent on whether given as treatment for bleeding episode or as prophylaxis
  Other Names: NNC 0129-0000-1003; N8-GP

SUMMARY:
This trial is conducted globally. The aim of the trial is to investigate the safety and efficacy of turoctocog alfa pegol (N8-GP) in previously untreated patients (PUPs) with haemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male, age below 6 years of age at the time of signing informed consent
* Diagnosis of severe haemophilia A (FVIII activity level 1%) based on medical records or central laboratory results
* No prior use of purified clotting factor products (5 previous exposures to blood components is acceptable)

Exclusion Criteria:

* Any history of FVIII inhibitor (defined by medical records) - Known or suspected hypersensitivity to trial product or related products
* Previous participation in this trial. Participation is defined as first dose administered of trial product
* Receipt of any investigational medicinal product within 30 days before screening
* Congenital or acquired coagulation disorder other than haemophilia A
* Any chronic disorder or severe disease which, in the opinion of the Investigator, might jeopardise the patient's safety or compliance with the protocol
* Patient's parent(s')/legally acceptable representative (LAR(s')) mental incapacity, unwillingness to cooperate, or a language barrier precluding adequate understanding and cooperation

Ages: 0 Years to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2014-06-26 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (95):
- United States (34):
  - Arizona H&T Phoenix Child Hosp, Phoenix, Arizona
  - Miller Children's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles - Endocrinology, Los Angeles, California
  - Children's Hosp Of Orange, Orange, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - Nemours Chld Clnc Jacksonville, Jacksonville, Florida
  - Nemours Child Orlando Hem/Onc, Orlando, Florida
  - St Joseph's Hospital Foundation, Tampa, Florida
  - Emory University_Atlanta_1, Atlanta, Georgia
  - Medical College Of Georgia, Augusta, Georgia
  - St. Luke's Mountain States Tumor Institute, Boise, Idaho
  - Rush University Med. Cntr, Chicago, Illinois
  - University Of Iowa, Iowa City, Iowa
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hosp-New Orleans, New Orleans, Louisiana
  - Univ of NE Med Center_Omaha, Omaha, Nebraska
  - Hemostasis and Thrombosis Center of Nevada, Las Vegas, Nevada
  - Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - The Brooklyn Hsptl Center, Brooklyn, New York
  - North Shore Long Island Jewish Medical Center, New Hyde Park, New York
  - Torrence Hemby Ped Hem/Onc Ctr, Charlotte, North Carolina
  - Novant Hlth Vasc Ins Charlotte, Charlotte, North Carolina
  - Univ Hosp Cleveland Med Ctr, Cleveland, Ohio
  - Dayton Children Hemostati Ctr, Dayton, Ohio
  - Univ Oklahoma Sci Ctr OK City, Oklahoma City, Oklahoma
  - Oregon Health & Science University_Portland_5, Portland, Oregon
  - Children's Hosptl Philadelphia, Philadelphia, Pennsylvania
  - St Christopher Hosp for Child, Philadelphia, Pennsylvania
  - Medical University Of SC, Charleston, South Carolina
  - Vanderbilt Hemostasis Thrombosis Clinic, Nashville, Tennessee
  - Univ of Utah Primary Children's Hospital, Salt Lake City, Utah
  - University Of Virginia Hospitl, Charlottesville, Virginia
  - Children's Hsptl Of The Kings, Norfolk, Virginia
- Algeria (2):
  - Beni Messous Hospital Issaad Hassani, Algiers
  - University Hospital Saadna Abdenour of Setif, Sétif
- Argentina (2):
  - Hospital de Pediatría S.A.M.I.C. "Prof. Dr. Juan P. Garrahan, CABA
  - Sanatorio Mayo Privado S.A, Córdoba
- Australia (2):
  - Lady Cilento Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
- Austria (7):
  - Med. Univ. Graz -Klinische Abteilung f. Allgemeine Pädiatrie, Graz
  - Universitätsklinik Kinder-Jugendheilkunde Innsbruck, Innsbruck
  - Klinikum Klagenfurt am Wörthersee (LKH Klagenfurt), Klagenfurt
  - Landes-Frauen und Kinderklinik Linz, Linz
  - LKH Salzburg- Univ. Klinik f. Kinder- und Jugendheilkunde, Salzburg
  - LKH St. Poelten, Kinder-und Jugendheilkunde, Sankt Pölten
  - Universitätsklinik für Kinder- und Jugendheilkunde, Vienna
- UMHAT Sveti Georgi EAD, Plovdiv, Clinic of Pediatrics, Plovdiv, Bulgaria
- Canada (2):
  - Health Science Centre, St. John's, Newfoundland and Labrador
  - Hamltn Hth Sci/McMstr Child Hosp, Hamilton, Ontario
- France (5):
  - Hospices Civils de Lyon- Hopital Louis Pradel-1, Bron
  - CHU Estaing, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Nantes-Hopital Hotel-Dieu, Nantes
  - Ap-Hp-Hopital Necker-1, Paris
  - Master centre for France, Paris La Défense
- Germany (4):
  - Coagulation Research Center, Duisburg
  - HZRM Haemophilie-Zentrum Rhein Main GmbH, Frankfurt am Main
  - Werlhof-Institut, Hanover
  - Universitätsklinikum des Saarlandes - Pädiatrische Onkologie und Hämatologie, Homburg/Saar
- Greece (2):
  - Aghia Sophia Childrens' Hospital, Athens
  - 'Ippokrateio' General Hospital of Thessaloniki, Thessaloniki
- Sheba MC - The Israeli National Hemophilia Center, Tel Litwinsky, Israel
- Italy (3):
  - Dipartimento di Ematologia Univ. Firenze, Florence
  - IRCCS Meyer Firenze, Florence
  - A.O.U. Città della Salute e della Scienza di Torino-Ospedale, Torino
- Japan (6):
  - Nagoya University Hospital_Blood Transfusion, Aichi
  - Hyogo prefectural kobe children's hospital, Hyōgo
  - Univ.HP, Kyoto Pref Univ of Medicine, Dept. of Pediatrics, Kyoto
  - Saitama Children's Med Centre_Hematology-Oncology, Saitama
  - Shizuoka Children's Hospital, Hematology-Oncology, Shizuoka
  - National Center for Child Health and Development_Hematology, Tokyo
- Malaysia (3):
  - Hospital Pulau Pinang_Georgetown, Penang, George Town, Pulau Pinang
  - Hospital Wanita dan Kanak-Kanak Kuala Lumpur, Kuala Lumpur
  - National Blood Centre, Kuala Lumpur
- Mexico (2):
  - Centro Medico Nacional SXXI-Hospital de Pediatria, IMSS, Mexico City, México, D.F.
  - Hospital Universitario Dr. José Eleuterio González_Monterrey, Monterrey, Nuevo León
- Portugal (2):
  - Centro Hospitalar Lisboa Norte-HSM, Lisbon
  - ULS São João, E.P.E., Porto
- Pediatric Hemophilia Program University, San Juan, Puerto Rico
- Romania (3):
  - ,,Louis Ţurcanu'' Emergency Hospital for Children, Timișoara, Timiș County
  - 1st Paediatric Department, Fundeni Clinical Institute, Bucharest
  - Emergency County Hospital Constanta, Constanța
- University Children's Hospital Tirsova, Belgrade, Serbia
- Spain (3):
  - Hospital Teresa Herrera Materno Infantil . E.O.X.I. A Coruña, A Coruña
  - Hospital Sant Joan de Déu, Esplugues Llobregat
  - Hospital Universitario La Paz, Madrid
- Taiwan (4):
  - Changhua Christian Hospital_Hematology Dept., Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital_Dept of Pediatrics, Kaohsiung City
  - China Medical University Children's Hospital, Taichung
  - National Taiwan University Children's Hospital, Taipei
- Thailand (3):
  - Sunpasitthiprasong Hospital_Pediatrics Department, Ubon Ratchathani, Mueang Distirct,
  - Ramathibodi Hospital_Paediatrics, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital _Pediatric Hematology and Oncology, Chiang Mai
- Ukraine (2):
  - SI Institute of Urgent and Recovery Surgery - Haematology, Donetsk
  - Institute of blood pathology and transfusion medicine of NAMSU - General and haematol. surgery, Lviv

REFERENCES:
- [Derived] Kenet G, Young G, Chuansumrit A, Matsushita T, Yadav V, Zak M, Male C. The immunogenicity, safety, and efficacy of N8-GP in previously untreated patients with severe hemophilia A: pathfinder6 end-of-trial results. J Thromb Haemost. 2023 Nov;21(11):3109-3116. doi: 10.1016/j.jtha.2023.07.030. Epub 2023 Aug 18. PMID 37597724
- [Derived] Male C, Konigs C, Dey S, Matsushita T, Millner AH, Zak M, Young G, Kenet G. The safety and efficacy of N8-GP (turoctocog alfa pegol) in previously untreated pediatric patients with hemophilia A. Blood Adv. 2023 Feb 28;7(4):620-629. doi: 10.1182/bloodadvances.2022007529. PMID 35858373
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 14 countries as follows: Australia (2), Austria (2), Bulgaria (1), Canada (1), Germany (1), Greece (2), Israel (1), Italy (1), Japan (3), Malaysia (3), Spain (2), Taiwan (1), Thailand (3), United States (8).
Pre-assignment Details: A total of 81 participants were exposed to Turoctocog alfa pegol (N8-GP). Trial consists of main phase: pre-prophylaxis, prophylaxis & immune tolerance induction (ITI) and extension phase: prophylaxis period until end of treatment. Pre-prophylaxis was optional and allowed participants to receive treatment until 24 months of age/upon reaching 20EDs, whichever came first. Other participants directly started on prophylaxis treatment at visit 1.
Groups:
- Pre-prophylaxis: At the beginning of the main phase of the trial, slow start prophylaxis and on-demand treatment of bleeding episodes with trial product (Turoctocog alfa pegol (N8-GP)) were allowed at the discretion of the investigator and participants parent(s)/ legally acceptable representative (LAR). The N8-GP dose for pre-prophylaxis treatment (except for bleeding episodes) was 60 International unit per kilogram (IU/kg) body weight (within the range of 50-75 IU/kg) to be administered as a single bolus dose intravenously (i.v.) with more than one week between doses (at the discretion of the investigator). Participants who developed FVIII inhibitors in the trial were shifted to ITI treatment.
- Prophylaxis: For prophylaxis treatment, regular N8-GP administration was initiated no later than at the participants age of 24 months, or after 20 EDs on pre-prophylaxis, whatever came first. During the main phase of the trial, participants received prophylaxis with i.v. injections of N8-GP preferably twice weekly, with doses separated by at least 3, and no more than 4, calendar days. Furthermore, it was permissible to start prophylaxis in the main phase with an every 3rd day or once-weekly dosing regimen. The N8-GP dose for prophylaxis treatment was 60 IU/kg (within the range of 50-75 IU/kg) to be administered as a single bolus dose i.v. on each administration day. Participants who developed FVIII inhibitors in the trial were shifted to ITI treatment.
- Immune Tolerance Induction (ITI): Participants who developed FVIII inhibitors in the trial were offered ITI treatment with N8-GP. If a newly diagnosed inhibitor participant still responded well to treatment with N8-GP, initiation of ITI could be postponed with up to 6 months, or ITI could be cancelled if the inhibitors had resolved during the 6 months. N8-GP treatment could continue in case of low titre FVIII inhibitor (lesser than or equal (≤) 5 Bethesda Units). In case of high titre FVIII inhibitor (greater than (>) 5 Bethesda Units), the investigator had to decide how to proceed with treatment. ITI with N8-GP had to be initiated within 6 months of the confirmatory inhibitor test. The N8-GP dose for ITI treatment was according to local standard. Maximum of 75 IU/kg as single dose, maximum of 200 IU/kg over 24 hours.
Period: Main Phase: Pre-Prophylaxis
Arm/Group | Pre-prophylaxis | Prophylaxis | Immune Tolerance Induction (ITI)
Started | 55 | 0 | 0
Completed | 44 | 0 | 0
Not Completed | 11 | 0 | 0
Not completed — Withdrawal by parent/guardian | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Other | 3 | 0 | 0
Period: Main Phase: Prophylaxis
Arm/Group | Pre-prophylaxis | Prophylaxis | Immune Tolerance Induction (ITI)
Started | 0 | 69 (44 participants were switched from pre-prophylaxis to other two groups during main phase (42 participants were switched to prophylaxis group and 2 participants were switched to immune tolerance induction (ITI) group). Out of 2 participants in immune tolerance induction (ITI) group, 1 participant was again switched from the ITI group to the prophylaxis group and additional 26 participants directly started the Prophylaxis period.) | 0
Completed | 0 | 55 | 0
Not Completed | 0 | 14 | 0
Not completed — Withdrawal by parent/guardian | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Adverse Event | 0 | 4 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Other | 0 | 1 | 0
Not completed — Switched to ITI without completing main phase | 0 | 2 | 0
Not completed — Early site closure | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Period: Immune Tolerance Induction
Arm/Group | Pre-prophylaxis | Prophylaxis | Immune Tolerance Induction (ITI)
Started | 0 | 0 | 8 (2 participants were switched from pre-prophylaxis and 6 participants were switched from prophylaxis to immune tolerance induction (ITI) group.)
Completed | 0 | 0 | 4
Not Completed | 0 | 0 | 4
Not completed — Withdrawal by parent/guardian | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Undergone minor surgery | 0 | 0 | 2
Period: Extension Phase: Prophylaxis
Arm/Group | Pre-prophylaxis | Prophylaxis | Immune Tolerance Induction (ITI)
Started | 0 | 55 | 0
Completed | 0 | 49 | 0
Not Completed | 0 | 6 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by parent/guardian | 0 | 1 | 0
Not completed — Other | 0 | 1 | 0
Not completed — Early site closure | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All participants that started the study.
Groups:
- All Participants: Participants received pre-prophylaxis treatment of N8-GP 60 IU/kg intravenous injection as slow start prophylaxis and on-demand treatment of bleeding episodes until they were 24 months of age or until 20 exposure days (ED) on pre-prophylaxis, whichever came first in the main phase. After which they switched to prophylaxis treatment. In prophylaxis, participants received N8-GP 60 IU/kg intravenous injection twice weekly with doses separated by at least 3, and no more than 4, calendar days. Furthermore, it was permissible to start prophylaxis in the main phase with an every 3rd day or once-weekly dosing regimen. In the extension phase, subjects were to continue the prophylaxis dosing regimen as prescribed at the end of the main phase.
Arm/Group | All Participants
Number analyzed (Participants) | 81
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 74
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 24
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 49
  More than one race | 0
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Inhibitory Antibodies Against Coagulation Factor VIII (FVIII)
Description: Number of participants with inhibitory antibodies against coagulation factor VIII (FVIII) was reported during the main and extension phase of the trial.
Time Frame: From start of the treatment up to 7 years
Population: Results were based on safety analysis set (SAS). The SAS consist of all participants exposed to N8-GP. Number of participants analyzed=participants with available data for this endpoint. This outcome is applicable only for the reported arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-prophylaxis | Prophylaxis
Number analyzed (Participants) | 55 | 68
Participants | 11 | 10

2. Secondary Outcome: Number of Adverse Events Including Serious Adverse Events and Medical Events of Special Interest
Description: Number of adverse events including serious adverse events and medical events of special interest reported during the main and extension phase of the trial. An adverse event (AE) is any untoward medical occurrence in a patient administered a product, and which does not necessarily have a causal relationship with this treatment. Serious adverse event (SAE) is an experience that at any dose results in any of the following: Death, a life-threatening experience, in-patient hospitalisation or prolongation of existing hospitalisation, persistent or significant disability or incapacity, congenital anomaly or birth defect and important medical events that may not result in death, be life threatening or require hospitalisation. Medical event of special interest (MESI) is an event which, in the evaluation of safety, has a special focus.
Time Frame: From start of the treatment up to 8.9 years
Population: Results were based on SAS. The SAS consists of all participants exposed to N8-GP.
Measure: Number; unit: Events
Arm/Group | Pre-prophylaxis | Prophylaxis | Immune Tolerance Induction (ITI)
Number analyzed (Participants) | 55 | 69 | 8
Events
  Adverse events | 116 | 644 | 32
  Serious adverse events | 24 | 56 | 3
  Medical events of special interest | 17 | 47 | 0

3. Secondary Outcome: Number of Participants With Confirmed High Titre Inhibitors (Defined as Inhibitor Titre Above 5 Bethesda Units (BU)
Description: Number of participants with confirmed high titre inhibitors (defined as inhibitor titre above 5 Bethesda Units (BU) was reported during the main and extension phase of the trial.
Time Frame: From start of the treatment up to 8.9 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-prophylaxis | Prophylaxis
Number analyzed (Participants) | 55 | 68
Participants | 3 | 8

4. Secondary Outcome: Number of Breakthrough Bleeding Episodes During Prophylaxis With N8-GP (Annualised Bleeding Rate)
Description: The number of bleeding episodes per year reported during the prophylactic treatment with N8-GP was reported.
Time Frame: From start of the treatment up to 8.9 years
Population: Results were based on full analysis set (FAS). The FAS consists of all participants exposed to N8-GP. The endpoint is applicable for only reported group. This outcome is applicable only for the reported arms.
Measure: Median (Inter-Quartile Range); unit: bleeds/patient/year
Arm/Group | Prophylaxis
Number analyzed (Participants) | 69
bleeds/patient/year | 1.35 [0.60 to 3.50]

5. Secondary Outcome: Haemostatic Effect of N8-GP in Treatment of Bleeding Episodes, Assessed by a Predefined 4-point Haemostatic Response Scale ("Excellent", "Good", "Moderate" and "None")
Description: Haemostatic effect of turoctocog alfa pegol for treatment of bleeding episodes was assessed by 4-point response scale: none, moderate, good or excellent. Excellent: Abrupt pain relief and/or clear improvement in objective signs of bleeding within approximately 8 hours after a single injection; Good: Definite pain relief and/or improvement in signs of bleeding within approximately 8 hours after a single injection, but possibly requiring more than one injection for complete resolution; Moderate: Probable or slight beneficial effect within approximately 8 hours after the first injection, but usually requiring more than one injection; None: No improvement, or worsening of symptoms. Number of bleeding episodes in each category is reported.
Time Frame: From start of the treatment up to 8.9 years
Population: Results were based on full analysis set (FAS). The FAS consists of all participants exposed to N8-GP. Number of participants analyzed=participants with available data for this endpoint.
Measure: Number; unit: Bleeding episodes
Units Other Than Participants: Bleeds
Arm/Group | Pre-prophylaxis | Prophylaxis | Immune Tolerance Induction (ITI)
Number analyzed (Participants) | 48 | 59 | 4
Number analyzed (Bleeds) | 160 | 345 | 8
Bleeding episodes
  Excellent | 69 | 227 | 2
  Good | 62 | 92 | 3
  Moderate | 18 | 18 | 3
  None | 3 | 6 | 0
  Missing | 8 | 2 | 0

6. Secondary Outcome: Consumption of N8-GP for Prophylaxis (International Unit Per Kilogram (IU/Kg))
Description: Consumption of N8-GP for prophylaxis is reported. Consumption used for treatment includes all doses given. Yearly consumption is only calculated for patients with a exposure time of at least 30 days. Average dose consumption in IU/kg during main and extension phase is reported.
Time Frame: From start of the treatment up to 8.9 years
Population: Results were based on full analysis set (FAS). The FAS consists of all participants exposed to N8-GP. The endpoint is applicable for only reported arm.
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | Prophylaxis
Number analyzed (Participants) | 69
IU/kg | 68.9 (7.6)

7. Secondary Outcome: Consumption of N8-GP for Prophylaxis (Number of Injections)
Description: Consumption of N8-GP for prophylaxis is reported. Consumption used for treatment includes all doses given. Yearly consumption is only calculated for patients with a exposure time of at least 30 days. Number of injections consumption per patient during main and extension phase is reported.
Time Frame: From start of the treatment up to 8.9 years
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Injections/patient
Arm/Group | Prophylaxis
Number analyzed (Participants) | 69
Injections/patient | 236.6 (208.2)

8. Secondary Outcome: Consumption of N8-GP for Treatment of Bleeding Episodes (International Unit Per Kilogram Per Bleed (IU/kg/Bleed))
Description: Consumption of N8-GP for treatment of bleeding episodes (IU/kg/bleed) is reported. Average dose consumption in IU/kg/bleed during main and extension phase is reported.
Time Frame: From start of the treatment up to 8.9 years
Population: Results were based on full analysis set (FAS). The FAS consists of all participants exposed to N8-GP. This outcome is applicable only for the reported arms.
Measure: Mean (Standard Deviation); unit: IU/kg/bleed
Arm/Group | Pre-prophylaxis | Prophylaxis
Number analyzed (Participants) | 55 | 69
IU/kg/bleed | 112.9 (113.4) | 92.1 (71.7)

9. Secondary Outcome: Consumption of N8-GP for Treatment of Bleeding Episodes (Number of Injections)
Description: Consumption of N8-GP for treatment of bleeding episodes (number of injections) is reported. Number of average injections required for treatment of per bleed is reported.
Time Frame: From start of the treatment up to 8.9 years
Population: Results were based on full analysis set (FAS). The FAS consists of all participants exposed to N8-GP.
Measure: Mean (Standard Deviation); unit: Injections/bleed
Arm/Group | Pre-prophylaxis | Prophylaxis
Number analyzed (Participants) | 55 | 69
Injections/bleed | 1.6 (1.6) | 1.3 (1.1)

10. Secondary Outcome: Total Consumption of N8-GP Per Patient (Prevention and Treatment of Bleeding Episodes) Annualised Value
Description: Total consumption of N8-GP per patient (prevention and treatment of bleeding episodes) annualised value is presented. Consumption used for treatment includes all doses given. Yearly consumption is only calculated for patients with a exposure time of at least 30 days. Consumption used for treatment per year per patient (IU/kg/year/patient) is reported.
Time Frame: From start of the treatment up to 8.9 years
Population: Results were based on full analysis set (FAS). The FAS consists of all participants exposed to N8-GP. Number of participants analyzed=participants with available data for this endpoint. This outcome is applicable only for the reported arms.
Measure: Mean (Standard Deviation); unit: IU/kg/year/patient
Arm/Group | Pre-prophylaxis | Prophylaxis
Number analyzed (Participants) | 50 | 69
IU/kg/year/patient | 2108.6 (2697.6) | 5394.9 (1887.9)

11. Secondary Outcome: Outcome of ITI, Assessed by a Predefined 4-point ITI Outcome Scale ("Success", "Partial Success", "Failure", "Other")
Description: The outcome of ITI was evaluated by predefined 4-point outcome of ITI scale ('success', 'partial success', 'failure', 'other'). Success: An inhibitor titre less than (<) 0.6 BU. A normalised FVIII recovery, defined as greater than or equal to (≥) 66 percentage (%) of expected incremental recovery. An N8-GP half-life (t½) ≥9 hours after a 72-hour treatment-free washout period. Partial success: Reduction in inhibitor titre to less than or equal to (≤) 5 BU. Clinical effect of N8-GP therapy as judged by the investigator. Failure: Failure to attain defined success or partial success within 24 months of uninterrupted ITI with N8-GP. Inhibitor decrease less than (<) 20% after one year of ITI treatment. Other: Not fulfilling the above criteria. Number of participants in each category is reported.
Time Frame: From start of the treatment up to 8.9 years
Population: Results were based on full analysis set (FAS). This outcome is applicable only for the reported arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Immune Tolerance Induction (ITI)
Number analyzed (Participants) | 8
Participants
  Success | 4
  Partial success | 2
  Failure | 2

ADVERSE EVENTS:
Time Frame: From start of the treatment up to 8.9 years
Description: All the presented adverse events (AEs) are treatment emergent adverse events (TEAEs). AEs occurring in a patient before being exposed to N8-GP. Safety analysis set included all patients exposed to N8-GP. Collective data for main and extension phase is reported for each group.
Arm/Group | Pre-prophylaxis | Prophylaxis | Immune Tolerance Induction (ITI)
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/69 | 0/8
Serious Adverse Events (participants affected / at risk) | 18/55 | 34/69 | 1/8
Other Adverse Events (participants affected / at risk) | 28/55 | 51/69 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-prophylaxis (N=55) | Prophylaxis (N=69) | Immune Tolerance Induction (ITI) (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Anti factor VIII antibody positive (Investigations) | 0 (0) | 2 (2) | 0 (0)
Arteriovenous fistula operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Device issue (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Enterobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Factor VIII inhibition (Blood and lymphatic system disorders) | 10 (10) | 12 (13) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Post procedural fistula (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Spinal epidural haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Therapy non-responder (General disorders) | 0 (0) | 1 (1) | 0 (0)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Urethral repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Urogenital fistula repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Vaccination site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-prophylaxis (N=55) | Prophylaxis (N=69) | Immune Tolerance Induction (ITI) (N=8)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 1 (2)
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Anti factor VIII antibody positive (Investigations) | 3 (3) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 6 (6) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 5 (6) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (5) | 5 (72) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (13) | 0 (0)
Cyanosis (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 6 (9) | 1 (1)
Ear infection (Infections and infestations) | 3 (7) | 9 (13) | 0 (0)
Factor VIII inhibition (Blood and lymphatic system disorders) | 0 (0) | 4 (6) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 9 (10) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 6 (7) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (7) | 22 (80) | 1 (5)
Otitis media (Infections and infestations) | 2 (2) | 4 (6) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 5 (8) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Pyrexia (General disorders) | 5 (6) | 26 (75) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 5 (10) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (13) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2) | 6 (8) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (3)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 16 (35) | 2 (3)
Varicella (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (10) | 1 (1)
Vaccine complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT02137850/Prot_SAP_000.pdf